CLINICAL TRIAL: NCT06814977
Title: Researching the Implementation of Acupuncture for Chronic Musculoskeletal Pain in Diverse Underserved Cancer Survivors (ReIMAGINE)
Brief Title: An Acupuncture Study for Cancer Survivors With Joint Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24-305
Record Dates: First submitted 2025-02-03; First posted 2025-02-07 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Cancer Survivor
Keywords: history of cancer; acupuncture; cancer; 24-305
MeSH Terms: conditions — Neoplasms | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acupuncture (Experimental): Participants will receive 10 weekly acupuncture treatments over 10 weeks.
  Interventions: Procedure: Acupuncture
- Usual Care (No Intervention): Participants will receive standard medical care, including pain medications and other treatments

INTERVENTIONS:
Procedure: Acupuncture — Acupuncture is a non-pharmacological intervention that does not involve the use of any therapeutic agents or devices. Participants will receive 10 weekly treatments over 10 weeks.
  Arms: Acupuncture

SUMMARY:
The purpose of this study is to see whether acupuncture is a practical (feasible) treatment for cancer survivors with joint pain.

ELIGIBILITY:
Inclusion Criteria:

* English- or Spanish-speaking adults
* Non white or Hispanic women with a prior cancer diagnosis
* Stable oncological disease or no evidence oncological of disease per clinical documentation or clinician assessment
* Worst pain rated ≥4 on a 0-10 scale in the preceding week
* ≥15 days with pain in the past 30 days
* Pain lasting ≥1 month
* Willing and able to complete questionnaires and other study activities
* Willing and able to provide informed consent for the trial

Exclusion Criteria:

* Completed active treatment (chemotherapy, surgery, radiation, transplantation) <4 weeks prior to study
* Maintenance therapies are allowed
* Pain attributed to inflammatory arthritis (e.g., rheumatoid arthritis, gout)
* Other non-musculoskeletal pain syndromes (eg, headache, visceral abdominal pain, neuropathic pain) can be present as comorbid conditions if the patient reports musculoskeletal pain as the primary source of pain
* Procedures involving affected joints within the last month or planned in the next 14 weeks
* Acupuncture use for pain in the past three months
* Implanted electronic device (e.g., pacemaker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Study feasibility as measured by rates of enrollment | 1 year
  The primary purpose of this study is to determine the feasibility of studying an acupuncture intervention for chronic musculoskeletal pain in racially/ethnically diverse, community-based cancer survivors.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Liou, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Memorial Sloan Kettering Cancer Center (All protocol activites), New York, New York
  - Jamaica Hospital Medical Center, Richmond Hill, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org